CLINICAL TRIAL: NCT00654706
Title: A Randomised, Double-Blind, Parallel-Group, Flexible-Dose Study Exploring the Neurocognitive Effect of Sertindole Versus Comparator in Patients With Schizophrenia Using the MATRICS Consensus Cognitive Battery (MCCB)
Brief Title: Efficacy Study Exploring the Effects on Cognition of Sertindole Versus Comparator in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11723A
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia; Cognition
Keywords: Schizophrenia; Cognition; MATRICS Consensus Cognitive Battery
MeSH Terms: conditions — Schizophrenia | interventions — sertindole; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertindole (Experimental)
  Interventions: Drug: Sertindole
- Quetiapine (Active Comparator)
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Sertindole — Once daily oral dose. Day 1-20: 4-16 mg/day (titration period). Day 21-84: 12, 16 or 20 mg/day (flexible treatment period).
  Arms: Sertindole
Drug: Quetiapine — Twice daily oral dose. Day 1-20: 50-500 mg/day (titration period). Day 21-84: 400, 500 or 600 mg/day (flexible treatment period).
  Arms: Quetiapine

SUMMARY:
The objective of this study is to explore the neurocognitive efficacy of Sertindole versus comparator in patients with schizophrenia using the MCCB.

DETAILED DESCRIPTION:
Sertindole is an atypical antipsychotic approved in the European Union (EU) for use in patients with schizophrenia who are intolerant to at least one other antipsychotic agent. During clinical development sertindole was found to be as effective in the treatment of schizophrenia as the first-generation antipsychotic haloperidol and as the second-generation antipsychotic risperidone.

Sertindole is generally well tolerated and has a benign side-effect profile, including an absence of sedation, no effect on plasma prolactin levels, moderate weight gain, no anticholinergic-mediated cognitive impairment and a low rate of extrapyramidal symptoms (EPS). Sertindole has been shown to prolong the QT interval and is contraindicated in patients with prolonged QT interval and in patients receiving drugs known to significantly prolong the QT interval.

The study is designed to provide data on the neurocognitive properties of sertindole versus quetiapine in patients with schizophrenia. Efficacy for cognitive impairment is assessed in patients who are in a stable phase of their illness, with a predefined maximum level of symptoms that will allow them to be included in the study. Prior antipsychotic medication will be withdrawn (down-tapered) and patients will be randomly assigned to one of the study drugs.

Cognitive deficiencies are an important feature of schizophrenia and correlate strongly with functional impairment. Improving functional outcomes in schizophrenia has a high priority and has resulted in the initiation of a program called Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) leading to the development of a neuropsychological test battery, the MCCB which is used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of schizophrenia
* Man or woman, aged between 18 and 55 years

Exclusion Criteria:

* Current Axis I primary psychiatric diagnosis other than schizophrenia
* Not previously received antipsychotic drugs for schizophrenia
* Acute exacerbation requiring hospitalisation within the last 3 months
* Clinically significant extrapyramidal symptoms
* Clinically significant cardiovascular disease, congestive heart failure, cardiac hypertrophy, arrhythmia or bradycardia
* Congenital long QT syndrome or a family history of this disease, or known acquired QT interval prolongation
* Significant ECG abnormalities
* Hypokalaemia or hypomagnesaemia
* In concurrent treatment with drugs inhibiting the P450 enzymes system CYP3A

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Neurocognitive effect of treatment based on the overall composite score on the MCCB | 12 weeks

SECONDARY OUTCOMES:
Domain specific scores on MCCB; PANSS total score, PANSS positive symptom subscale score, PANSS negative symptom subscale score, and PANSS general psychopathology subscale score; CGI-S, CDSS and GAF scores; QLS and UPSA total and subscale scores; ECGs | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (26):
- United States (26):
  - US017, Garden Grove, California
  - US008, National City, California
  - US001, Pasadena, California
  - US006, Pico Rivera, California
  - US011, San Diego, California
  - US014, Stanford, California
  - US026, Torrance, California
  - US016, Aurora, Colorado
  - US015, Orange City, Florida
  - US010, Tampa, Florida
  - US007, Atlanta, Georgia
  - US024, Chicago, Illinois
  - US002, Joliet, Illinois
  - US012, Baltimore, Maryland
  - US027, Glen Burnie, Maryland
  - US019, Lebanon, New Hampshire
  - US021, Clementon, New Jersey
  - US013, Brooklyn, New York
  - US025, Staten Island, New York
  - US005, Charlotte, North Carolina
  - US018, Durham, North Carolina
  - US022, Philadelphia, Pennsylvania
  - US023, Austin, Texas
  - US020, Dallas, Texas
  - US004, DeSoto, Texas
  - US028, Houston, Texas

REFERENCES:
- [Derived] Nielsen J, Matz J, Mittoux A, Polcwiartek C, Struijk JJ, Toft E, Kanters JK, Graff C. Cardiac effects of sertindole and quetiapine: analysis of ECGs from a randomized double-blind study in patients with schizophrenia. Eur Neuropsychopharmacol. 2015 Mar;25(3):303-11. doi: 10.1016/j.euroneuro.2014.12.005. Epub 2015 Jan 3. PMID 25583364